CLINICAL TRIAL: NCT02551237
Title: A Phase III Study Evaluating Two Neoadjuvant Treatments Radiochemotherapy (5 Weeks - 50Gy+Capecitabine) and Radiotherapy (1week - 25Gy) in Patient Over 75 With Locally Advanced Rectal Carcinoma
Brief Title: Neoadjuvant Treatment for Advanced Rectal Carcinoma
Acronym: NACRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 42 GERICO12/UCGI; 2015-A01365-44 (Other: ID-RCB); UC-0103/1503 (Other: UNICANCER)
Record Dates: First submitted 2015-08-31; First posted 2015-09-16 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Rectal Carcinoma
Keywords: Elderly patient; Radiotherapy; Radio chemotherapy; Neoadjuvant treatment
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiochemotherapy (Active Comparator): Patients who will be treated with
  * radiotherapy 50 Gy in 25 fractions of 2 Gy, five times per week, over a period of 5 weeks associated with
  * oral capecitabine 800 mg/m2 twice daily from the first day of radiotherapy and given 5 days per week during radiotherapy.
  The surgery will be planned 7 weeks (±1 week) after the end of preoperative treatment
  Interventions: Radiation: 50 Gy; Drug: Capecitabine
- Radiotherapy (Experimental): Patients who will be treated with radiotherapy 25 Gy in 5 fractions of 5 Gy delivered in one week (short-course arm) without chemotherapy.
  The surgery will be planned 7 weeks (±1 week) after the end of preoperative treatment
  Interventions: Radiation: 25 Gy

INTERVENTIONS:
Radiation: 50 Gy — radiotherapy 50 Gy in 25 fractions of 2 Gy, five times per week, over a period of 5 weeks
  Arms: Radiochemotherapy
Drug: Capecitabine — oral capecitabine 800 mg/m2 twice daily from the first day of radiotherapy and given 5 days per week during radiotherapy.
  Other Names: Xeloda
  Arms: Radiochemotherapy
Radiation: 25 Gy — radiotherapy 25 Gy in 5 fractions of 5 Gy delivered in one week (short-course arm)
  Arms: Radiotherapy

SUMMARY:
The purpose of the study is to compare pre-operative radio-chemotherapy (RT + capecitabine) to a short course RT associated with a delayed surgery, with two primary objectives: the efficacy evaluation (rate of R0 resection) and the preservation of autonomy (score IADL).

DETAILED DESCRIPTION:
Colorectal cancer is one of the most frequent cancers diagnosed in France. The average age of diagnosis in 2012 was 70 years old for men and 73 years for women, confirming that colorectal cancer is a disease of the elderly population.

The literature concerning combined treatments of colorectal cancer in the elderly is extremely limited. The application of combined treatments in the geriatric population is associated with an increase in the therapeutic complications. These post-operative complications together with the comorbidities and age are unfavorable prognostic factors for survival in patients with cancer of the rectum; this explains why the improved results obtained during the last decades are perceptible in younger patients and not in the elderly.

In the general population, pre-operative radio-chemotherapy has imposed itself as a standard treatment for the cancer of the rectum locally advanced. The utilization of fluoropyrimidines associated with radiotherapy (RT) delivered in fractions [long course RT (50 Gy in 5 weeks), surgery planned 6 to 8 weeks later] increases the complete histological response rate and decreases significantly the rate of local relapse.

The short-course RT [short course RT using the Swedish model (5x5 Gy in 5 days), with the surgery programmed the following week] is the standard neoadjuvant protocol in an important number of countries and/or academic groups. The studies that have compared the fractioned RT scheme to the short-course RT protocols have not shown any evidence of a change in efficacy of the short course RT concerning the following criteria: rate of R0 resection, rate of sphincter conservation, rate of relapse at 3 years, the disease free survival or the overall survival. Similarly, there appears to be no difference in severe toxicities in the long term. It should however be noted that short-course RT followed by immediate surgery may be less efficient than combined treatment in patients with a distal T3 cancer, even though these conclusions published by Ngan have been criticized by certain. On the other hand, the fractioned combined treatments results in more tumor and stage reduction and thus more sterilization.

Nevertheless a retrospective analysis, performed in the Stockholm region, in patients irradiated with short-course protocol but operated with a delay of at least 4 weeks resulted in a sterilization rate of 8%. This result is even more interesting since in this cohort, 46% of the patients had a tumor classified T4 and that 38% of the patients had a primitive tumor considered inoperable.

In the elderly population, the neoadjuvant treatment has rarely been studied. An exploratory analysis of the PRODIGE 2 study, based on age as the criteria, has shown that pre-operative radio-chemotherapy is significantly more toxic in the elderly population, from 70 years of age. Globally the lower tolerance for the pre-operative radio-chemotherapy results in more frequent early termination of RT and a statistically significant decrease in the number of patients operated. Furthermore, if the type of surgery was not significantly different between patients <70 years and those ≥70 years, we observe a non-significant increase in the rate of prolonged stoma (patients amputated without closure of the stoma). These differences in the surgical procedures is also observed in other publications, placing the emphasis on the fact that in the absence of any difference in the clinical presentation or the characteristic of the tumor, the risk of real or supposed decompensation modifies the surgical care. These data, as well as those in the literature, provides evidence that the pre-operative radio-chemotherapy strategy followed by surgery, the standard strategy in younger patients, is associated with more side effects in the elderly, resulting in the benefit-risk balance, in this population, to be more questionable.

It is therefore necessary to conduct a specific studies in the elderly population, with cancer of the rectum with the objective to maintain the carcinological results obtained with classical radio-chemotherapy with at the same time better controlling the secondary effects of the treatment and the risk of decompensation of the patients: the short course radiotherapy associated with a delayed surgery may be a therapeutic scheme well adapted to this population.

The investigators therefore propose a study comparing pre-operative radio-chemotherapy (RT + capecitabine) to a short course RT associated with a delayed surgery, with two primary objectives: the efficacy evaluation (rate of R0 resection) and the preservation of autonomy (score IADL).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥75 years
* Eastern Cooperative Oncology Group (ECOG) ≤2
* Adenocarcinoma of the rectum histologically proven
* Tumor ≤12 cm from the anal margin, the measurement done by rigid rectoscopy or by sub peritoneal MRI
* Require a pre-operative treatment (tumor classified T3 or T4 resectable by MRI and tomodensitometry or T2 of the very low rectum)
* Patient operable
* No radiologically detectable metastases
* Absolute Neutrophile count (ANC) ≥1500/mm³; Platelets ≥100 000/mm³ and Hemoglobin ≥10 g/dL
* Bilirubin ≤1.5 x upper limit of normal (ULN), aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤1.5 x upper limit of normal (ULN), Alkaline Phosphatase ≤1.5 x upper limit of normal (ULN)
* Creatinine clearance ≥30 ml/min (Cockcroft and Gault)
* Uracilemia < 16ng/mL
* Public or private Health Insurance coverage
* Patient has been informed and signed the informed consent document

Exclusion Criteria:

* Non-resectable tumor
* History of chronic diarrhea or an inflammatory disease of the colon or rectum, or intestinal obstruction or sub-obstruction
* History of pelvic radiotherapy
* Any active febrile infection or any other serious underlying pathology that may prevent the patient from receiving the treatment
* Significant Cardiovascular diseases such as, but not limited to: cardiovascular or myocardial infarction ≤6 months before inclusion, congestive heart failure class II or higher (NYHA), unstable angina, arrhythmia requiring medication or uncontrolled hypertension;
* Significative cardiovascular conditions such as, but not limited to : Cardiac angioplasty or stenting, Myocardial infarction, Unstable angina, Coronary artery bypass graft surgery Symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA), clinically significant irregular heartbeat requiring medication
* Severe and unexpected reactions to fluoropyrimidine therapy
* Any contra-indication to capecitabine and its excipients; patients with hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not included.
* Uracilemia ≥ 16ng/mL
* Any other concomitant cancer or history of cancer in the last 3 years, with the exception of the in situ cancer of the uterus, treated, or squamous-cell or basal-cell carcinoma.
* Patients already included in another therapeutic trail with an experimental molecule
* Person deprived of liberty
* Patient that for geographical, social and/or physical reasons will not be able to follow the procedure as required by the protocol

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 3 months
  Compare the efficacy between the arm A and the arm B (with an objective of non-inferiority)
IADL (Instrumental Activities of Daily Living) Score | 1 year
  Compare the maintenance of autonomy between the arm A and arm B (with an objective of superiority)

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.03 | 3 months
  Description of the Adverse Events during the pre-operative period.
Post-operative complications | 3 months
  according to Dindo-Clavien classification
Death rate | at 6 and 12 months
  Death rate is defined as the percentage of patients who died since the date of randomisation at 6 and 12 months post-surgery (M6 and M12) from any cause
Overall survival (OS) | 10 years
  The OS is defined as the interval between the date of randomization and the date of deaths from any cause
Specific survival | 10 years
  The specific survival is defined as the interval between the date of randomization and the date of deaths due to cancer.
Disease free survival | 10 years
  The disease free survival is defined as the interval between the date of randomization and the date of cancer relapse (local regional or distant), second cancer or death from any cause.
Loco-regional disease free survival | 10 years
  The disease free survival is defined as the interval between the date of randomization and the date of cancer relapse (local or regional).
Rate of stoma | at 6 and 12 months
  percentage of patients with definitive or transitional stoma after surgery.
Instrumental Activities of Daily Living (IADL) | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Autonomy Assessment
Activities of Daily Living (ADL) | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Autonomy Assessment
Questionnaire G8 | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Geriatric Screening
Mini-Mental Score Examination (MMSE) | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Cognitive functioning
Walking gate | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
Geriatric Depression Scale (GDS15) | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Depression Assessment
Charlson score | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Comorbidities evaluation
Mini Nutritional Assessment (MNA) | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Nutritional Evaluation
EORTC QLQ-C30 + EDL14 | Baseline, within 2 weeks before surgery and 3, 6 and 12 months after surgery
  Quality of Life (QLQ)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Francois, Principal Investigator — Centre Antoine Lacassagne
Locations (37):
- France (37):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Clinique Claude Bernard, Albi
  - CHU Amiens Picardie, Amiens
  - Polyclinique Maymard, Bastia
  - Centre Hospitalier de Beauvais, Beauvais
  - CHU de Besançon, Besançon
  - Cebtre Hospitalier de Blois, Blois
  - Hôpital Avicenne, Bobigny
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - CHU Henri Mondor, Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre Georges François Leclerc, Dijon
  - CHU DIJON (Hôpital du Bocage), Dijon
  - CHIC des Alpes du Sud- site de Gap, Gap
  - CHU de Grenoble Hôpital A Michallon, Grenoble
  - Hôpital Privé Sainte Marguerite, Hyères
  - CHD de Vendée, La Roche-sur-Yon
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - CHU Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Centre azuréen de cancérologie, Mougins
  - Hôpital Américain de Paris, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Centre Médical Oncogard Institut de cancérologie du Gard, Nîmes
  - Chu Caremeau, Nîmes
  - Hôpital TENON, Paris
  - CHU de Bordeaux, Pessac
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Henri Becquerel, Rouen
  - Hôpital d'instruction des Armées, Saint-Mandé
  - Clinique Pasteur, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus Grand Paris, Villejuif

REFERENCES:
- [Derived] Francois E, De Bari B, Ronchin P, Nouhaud E, Martel-Lafay I, Artru P, Clavere P, Vendrely V, Boige V, Gargot D, Lemanski C, De Sousa Carvalho N, Gal J, Pernot M, Magne N. Comparison of short course radiotherapy with chemoradiotherapy for locally advanced rectal cancers in the elderly: A multicentre, randomised, non-blinded, phase 3 trial. Eur J Cancer. 2023 Feb;180:62-70. doi: 10.1016/j.ejca.2022.11.020. Epub 2022 Nov 28. PMID 36535196